CLINICAL TRIAL: NCT03142334
Title: A Phase 3, Randomized, Double-Blind, Placebo-Controlled Clinical Trial of Pembrolizumab (MK-3475) as Monotherapy in the Adjuvant Treatment of Renal Cell Carcinoma Post Nephrectomy (KEYNOTE-564)
Brief Title: Safety and Efficacy Study of Pembrolizumab (MK-3475) as Monotherapy in the Adjuvant Treatment of Renal Cell Carcinoma Post Nephrectomy (MK-3475-564/KEYNOTE-564)
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 3475-564; 173704 (Registry Identifier: JAPAC-CTI); MK-3475-564 (Other: MSD); KEYNOTE-564 (Other: MSD); U1111-1275-8289 (Other: UTN); 2016-004351-75 (EudraCT Number)
Record Dates: First submitted 2017-05-03; First posted 2017-05-05 (Actual); Results first posted 2021-12-28 (Actual); Last update posted 2024-11-13 (Actual); Status verified 2024-11

CONDITIONS: Renal Cell Carcinoma
Keywords: Programmed Cell Death-1 (PD1, PD-1); Programmed Death-Ligand 1 (PDL1, PD-L1); Adjuvant
MeSH Terms: conditions — Carcinoma, Renal Cell; Parkinson Disease 4, Autosomal Dominant Lewy Body | interventions — pembrolizumab; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Pembrolizumab (Experimental): Participants receive pembrolizumab 200 mg via intravenous (IV) infusion on Day 1 of each 3-week cycle for up to 17 cycles (up to approximately 1 year).
  Interventions: Biological: Pembrolizumab
- Placebo (Placebo Comparator): Participants receive placebo (saline solution) via IV infusion on Day 1 of each 3-week cycle for up to 17 cycles (up to approximately 1 year).
  Interventions: Drug: Placebo

INTERVENTIONS:
Biological: Pembrolizumab — IV infusion
  Other Names: MK-3475; KEYTRUDA®; SCH 900475
  Arms: Pembrolizumab
Drug: Placebo — IV infusion
  Other Names: saline solution
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of pembrolizumab (MK-3475) in the adjuvant treatment of adult participants who have undergone nephrectomy and have intermediate-high risk, high risk, or M1 no evidence of disease (M1 NED) renal cell carcinoma (RCC) with clear cell component.

The primary study hypothesis is that pembrolizumab is superior to placebo with respect to Disease-free Survival (DFS) as assessed by the Investigator in male and female participants with intermediate-high risk, high risk and M1 NED RCC.

DETAILED DESCRIPTION:
Participants will be assigned to receive study treatment until disease recurrence, unacceptable adverse events (AEs), intercurrent illness that prevents further administration of treatment, Investigator's decision to withdraw the participant, noncompliance with study treatment or procedural requirements, administrative reasons requiring cessation of treatment, or until the participant has received 17 cycles of study treatment (approximately 1 year). Each cycle is 3 weeks long.

With Protocol Amendment 02 (dated 04 Sep 2019), the secondary study objectives for the evaluation of pharmacokinetic (PK) parameters and the presence of pembrolizumab antidrug antibodies (ADA) were reclassified as tertiary study objectives.

ELIGIBILITY:
Inclusion Criteria:

* Has histologically confirmed diagnosis of renal cell carcinoma (RCC) with clear cell component with or without sarcomatoid features
* Female participants of childbearing potential must be willing to use an adequate method of contraception, for the course of the study through 120 days after the last dose of study treatment
* Male participants of childbearing potential must agree to use an adequate method of contraception, starting with the first dose of study treatment through 120 days after the last dose of study treatment
* Has intermediate-high risk, high risk, or M1 no evidence of disease (NED) RCC as defined by the following pathological tumor-node-metastasis and Fuhrman grading status:

  1. Intermediate-high risk RCC: pT2, Grade 4 or sarcomatoid, N0, M0; pT3, Any Grade, N0, M0
  2. High risk RCC: pT4, Any Grade N0, M0; pT Any stage, Any Grade, N+, M0
  3. M1 NED RCC participants who present not only with the primary kidney tumor but also solid, isolated, soft tissue metastases that can be completely resected at one of the following: the time of nephrectomy (synchronous) or, ≤1 year from nephrectomy (metachronous)
* Has received no prior systemic therapy for advanced RCC
* Has undergone a partial nephroprotective or radical complete nephrectomy (and complete resection of solid, isolated, soft tissue metastatic lesion(s) in M1 NED participants) with negative surgical margins
* Must have undergone a nephrectomy and/or metastasectomy ≥28 days prior to signing informed consent and ≤12 weeks prior to randomization
* Must be tumor-free as assessed by the Investigator and validated by either computed tomography (CT) or magnetic resonance imaging (MRI) scan of the brain and chest, abdomen, and pelvis and a bone scan ≤28 days from randomization
* Must have provided adequate tissue per the following: Nephrectomy only: tissue from nephrectomy (required); Synchronous M1 NED: tissue from nephrectomy (required) AND, metastasectomy tissue (if available); Metachronous M1 NED: tissue from metastasectomy (required) AND, nephrectomy tissue (if available)
* Has an Eastern Cooperative Oncology Group Performance Status (ECOG PS) score of 0 or 1
* Has adequate organ function

Exclusion Criteria:

* Has had major surgery, other than nephrectomy and/or resection of pre-existing metastases for M1 NED participants, within 12 weeks prior to randomization
* Has received prior radiotherapy for RCC
* Has pre-existing brain or bone metastatic lesions
* Has residual thrombus post nephrectomy in the vena renalis or vena cava
* Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior the first dose of study treatment
* Has an active autoimmune disease that has required systemic treatment in past 2 years (i.e., with use of disease modifying agents, corticosteroids, or immunosuppressive drugs). Replacement therapy is allowed
* Has a known additional malignancy that is progressing or required active treatment ≤3 years ago. Exceptions include early-stage cancers (carcinoma in situ or Stage 1) treated with curative intent, basal cell carcinoma of the skin, squamous cell carcinoma of the skin, in situ cervical cancer, in situ prostate cancer, or in situ breast cancer that has undergone potentially curative therapy
* Has a history of (non-infectious) pneumonitis that required steroids or has current pneumonitis
* Has an active infection requiring systemic therapy
* Has a history of, or is currently on, dialysis
* Has a known history of human immunodeficiency virus (HIV) infection
* Has known active hepatitis B or hepatitis C virus infection
* Has a known history of active tuberculosis (Bacillus tuberculosis)
* Has had a prior solid organ transplant
* Has severe hypersensitivity (≥ Grade 3) to pembrolizumab and/or any of its excipients
* Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the study, starting with the Screening visit through 120 days after the last dose of study treatment
* Has received prior therapy with an anti-programmed cell death protein 1 (anti-PD-1), anti-programmed cell death-ligand 1 (anti-PD-L1), or anti-programmed cell death-ligand 2 (anti-PD-L2) agent or with an agent directed to another co-inhibitory T-cell receptor (i.e., cytotoxic T-lymphocyte-associated protein 4 [CTLA-4], OX-40, CD137 [tumor necrosis factor receptor superfamily member 9 (TNFRSF9)]) or has previously participated in a Merck pembrolizumab (MK-3475) clinical trial
* Has received prior anticancer therapy, monoclonal antibody, chemotherapy, or an investigational agent or device within 4 weeks or 5 half-lives (whichever is longer) before first dose of study treatment or not recovered (i.e., must be ≤ Grade 1 or at Baseline) from AEs due to previously administered agents
* Has received a live vaccine within 30 days prior to the first dose of study treatment
* Is currently participating in or has participated in a study of an investigational agent or has used an investigational device within 4 weeks prior to the first dose of study treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 994 (Actual)
Dates: Start 2017-06-09 (Actual); Primary Completion 2020-12-14 (Actual); Study Completion 2025-12-28 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (251):
- United States (62):
  - Arizona Oncology Associates, PC- HAL ( Site 8018), Phoenix, Arizona
  - USC Norris Comprehensive Cancer Center ( Site 0038), Los Angeles, California
  - UCSF Helen Diller Family Comprehensive Cancer Center ( Site 0056), San Francisco, California
  - Sansum Clinic Research ( Site 8014), Santa Barbara, California
  - Stanford Cancer Center ( Site 0028), Stanford, California
  - Rocky Mountain Cancer Center ( Site 8010), Aurora, Colorado
  - Georgetown University Medical Center ( Site 0002), Washington D.C., District of Columbia
  - Boca Raton Regional Hospital- Lynn Cancer Institute ( Site 0035), Boca Raton, Florida
  - Manatee Medical Research Institute ( Site 0039), Bradenton, Florida
  - Woodlands Medical Specialists, PA ( Site 8021), Pensacola, Florida
  - Northwest Georgia Oncology Centers PC ( Site 0014), Marietta, Georgia
  - Illinois Cancer Specialists ( Site 8001), Niles, Illinois
  - McFarland Clinic ( Site 0025), Ames, Iowa
  - University of Iowa Hospital and Clinics ( Site 0031), Iowa City, Iowa
  - University Medical Center New Orleans ( Site 0053), New Orleans, Louisiana
  - Weinberg Cancer Institute at Franklin Square ( Site 0046), Baltimore, Maryland
  - Maryland Oncology Hematology, P.A. ( Site 8020), Rockville, Maryland
  - Beth Israel Deaconess Medical Ctr. ( Site 0044), Boston, Massachusetts
  - Dana-Farber Cancer Institute (Boston) ( Site 0007), Boston, Massachusetts
  - University of Michigan ( Site 0045), Ann Arbor, Michigan
  - Karmanos Cancer Institute ( Site 0013), Detroit, Michigan
  - Henry Ford Hospital ( Site 0032), Detroit, Michigan
  - Quest Research Institute ( Site 0036), Royal Oak, Michigan
  - Fairview Southdale Medical Oncology Clinic ( Site 0041), Edina, Minnesota
  - Minnesota Oncology Specialist, PA ( Site 8002), Minneapolis, Minnesota
  - Park Nicollet Frauenshuh Cancer Center ( Site 0020), Saint Louis Park, Minnesota
  - St. Vincent Healthcare Frontier Cancer Center ( Site 0008), Billings, Montana
  - Nebraska Cancer Specialists ( Site 0012), Omaha, Nebraska
  - Comprehensive Cancer Centers of Nevada ( Site 8013), Las Vegas, Nevada
  - Rutgers Cancer Institute of New Jersey ( Site 0059), New Brunswick, New Jersey
  - University of New Mexico Cancer Center ( Site 0043), Albuquerque, New Mexico
  - Montefiore Medical Center ( Site 0009), The Bronx, New York
  - Duke University ( Site 0037), Durham, North Carolina
  - Oncology Hematology Care, Inc. ( Site 8008), Cincinnati, Ohio
  - Oklahoma Cancer Specialists and Research Institute, LLC ( Site 0052), Tulsa, Oklahoma
  - Northwest Cancer Specialists, P.C. ( Site 8006), Tigard, Oregon
  - St. Luke's University Health Network ( Site 0042), Easton, Pennsylvania
  - Abramson Cancer Center ( Site 0010), Philadelphia, Pennsylvania
  - Charleston Hematology Oncology Associates PA ( Site 8000), Charleston, South Carolina
  - Medical University of South Carolina ( Site 0033), Charleston, South Carolina
  - Avera Cancer Institute ( Site 0023), Sioux Falls, South Dakota
  - Urology Associates [Nashville, TN] ( Site 0063), Nashville, Tennessee
  - Texas Oncology-Austin Central ( Site 8003), Austin, Texas
  - Baylor Sammons Cancer Center/ Texas Oncology ( Site 8019), Dallas, Texas
  - UT Southwestern Medical Center ( Site 0003), Dallas, Texas
  - Texas Oncology-Denton South ( Site 8016), Denton, Texas
  - Texas Oncology-Memorial City ( Site 8015), Houston, Texas
  - MD Anderson Cancer Center ( Site 0065), Houston, Texas
  - UTHealth/Memorial Hermann Cancer Center ( Site 0001), Houston, Texas
  - Texas Oncology- Paris ( Site 8004), Paris, Texas
  - CTRC at The University of Texas Health Science Center at San Antonio ( Site 0026), San Antonio, Texas
  - Texas Oncology-Tyler ( Site 8005), Tyler, Texas
  - Texas Oncology-Waco ( Site 8012), Waco, Texas
  - IHO Corporation- Utah Cancer Specialists ( Site 0055), Salt Lake City, Utah
  - Virginia Oncology Associates ( Site 8011), Norfolk, Virginia
  - Providence Regional Cancer Partnership ( Site 0016), Everett, Washington
  - SCCA/UW ( Site 0029), Seattle, Washington
  - Cancer Care Northwest ( Site 0021), Spokane, Washington
  - Medical Oncology Associates (Summit Cancer Centers) ( Site 0005), Spokane, Washington
  - Northwest Medical Specialties, PLLC ( Site 0034), Tacoma, Washington
  - Yakima Valley Memorial Hospital North Star Lodge ( Site 8017), Yakima, Washington
  - University of Wisconsin Carbone Cancer Center ( Site 0019), Madison, Wisconsin
- Argentina (10):
  - Centro de Investigaciones Clinicas - Clinica Viedma ( Site 1102), Viedma, Río Negro Province
  - Sanatorio Parque ( Site 1104), Rosario, Santa Fe Province
  - Instituto de Investigaciones Metabolicas -I.D.I.M.- ( Site 1113), Buenos Aires
  - Fundacion Favaloro ( Site 1110), Buenos Aires
  - Instituto Medico Alexander Fleming ( Site 1105), Buenos Aires
  - Centro Oncologico Riojano Integral ( Site 1101), La Rioja
  - Centro Oncologico de Integracion Regional. COIR ( Site 1109), Mendoza
  - Sanatorio Britanico ( Site 1106), Rosario
  - Instituto de Oncologia de Rosario ( Site 1100), Rosario
  - Centro Medico San Roque ( Site 1108), San Miguel de Tucumán
- Australia (7):
  - Saint George Hospital [Kogarah, Australia] ( Site 0707), Kogarah, New South Wales
  - Macquarie University Hospital ( Site 0700), Macquarie Park, New South Wales
  - Adelaide Cancer Centre ( Site 0703), Kurralta Park, South Australia
  - Bendigo Cancer Centre ( Site 0704), Bendigo, Victoria
  - Box Hill Hospital ( Site 0701), Box Hill, Victoria
  - Fiona Stanley Hospital ( Site 0702), Murdoch, Western Australia
  - Ballarat Health Services ( Site 0705), Ballarat
- Brazil (12):
  - Instituto de Cancer e Transplante de Curitiba ICTR ( Site 1012), Curitiba, Paraná
  - Liga Norte Riograndense Contra o Cancer ( Site 1013), Natal, Rio Grande do Norte
  - Universidade de Caxias do Sul ( Site 1004), Caxias do Sul, Rio Grande do Sul
  - Hospital Bruno Born ( Site 1015), Lajeado, Rio Grande do Sul
  - Uniao Brasileira de Educacao e Assistencia Hospital Sao Lucas da Pucrs ( Site 1001), Porto Alegre, Rio Grande do Sul
  - Hospital Nossa Senhora da Conceicao ( Site 1000), Porto Alegre, Rio Grande do Sul
  - Fundacao Pio XII - Hospital de Cancer de Barretos ( Site 1002), Barretos, São Paulo
  - Fundacao Dr Amaral Carvalho ( Site 1005), Jaú, São Paulo
  - Instituto do Cancer de Sao Paulo - ICESP ( Site 1010), São Paulo, São Paulo
  - Casa de Saude Santa Marcelina ( Site 1006), São Paulo, São Paulo
  - Hosp. Clinicas da Fac. de Medicina de Ribeirao Preto - USP ( Site 1016), Ribeirão Preto
  - COT Centro Oncologico do Triangulo Ltda ( Site 1014), Uberlândia
- Canada (13):
  - CancerCare Manitoba ( Site 0119), Winnipeg, Manitoba
  - Dr. Leon Richard Oncology Centre ( Site 0106), Moncton, New Brunswick
  - William Osler Health System ( Site 0115), Brampton, Ontario
  - Juravinski Cancer Centre ( Site 0117), Hamilton, Ontario
  - London Regional Cancer Program - London HSC ( Site 0107), London, Ontario
  - Lakeridge Health ( Site 0108), Oshawa, Ontario
  - Niagara Health System - St. Catharines ( Site 0120), St. Catharines, Ontario
  - CIUSSS du Saguenay-Lac-St-Jean ( Site 0113), Chicoutimi, Quebec
  - CISSS-CA Hotel Dieu de Levis ( Site 0111), Lévis, Quebec
  - CIUSSS de l Est de L Ile de Montreal - Hopital Maisonneuve-Rosemont ( Site 0118), Montreal, Quebec
  - St-Jerome Medical Research Inc ( Site 0103), Saint-Jérôme, Quebec
  - Allan Blair Cancer Centre ( Site 0116), Regina, Saskatchewan
  - Saskatoon Cancer Centre ( Site 0105), Saskatoon, Saskatchewan
- Chile (12):
  - Instituto Nacional del Cancer ( Site 0912), Santiago, Santiago Metropolitan
  - Centro Oncologico Antofagasta ( Site 0914), Antofagasta
  - Hospital Regional de La Serena ( Site 0907), La Serena
  - Hospital Regional Rancagua Libertador Bernardo O Higgins ( Site 0910), Rancagua
  - Health and Care Chile ( Site 0901), Santiago
  - Fundacion Arturo Lopez Perez FALP ( Site 0902), Santiago
  - Iram Cancer Research ( Site 0909), Santiago
  - Hospital Militar de Santiago ( Site 0911), Santiago
  - Pontificia Universidad Catolica de Chile ( Site 0904), Santiago
  - Hospital Clinico Universidad de Chile ( Site 0905), Santiago
  - Sociedad de Investigaciones Medicas Limitadas ( Site 0913), Temuco
  - Oncocentro ( Site 0900), Viña del Mar
- Colombia (8):
  - Hospital Pablo Tobon Uribe. ( Site 0805), Medellín, Antioquia
  - Clinica de la Costa Ltda. ( Site 0804), Barranquilla, Atlántico
  - Sociedad de Hematologia y Oncologia del Cesar ( Site 0809), Valledupar, Cesar Department
  - Instituto Nacional de Cancerologia E.S.E ( Site 0807), Bogota, Cundinamarca
  - Oncologos del Occidente S.A. ( Site 0800), Pereira, Risaralda Department
  - Fundacion CardioInfantil Instituto de Cardiologia ( Site 0803), Bogotá
  - Administradora Country SA - Clinica del Country ( Site 0808), Bogotá
  - Oncomedica S.A. ( Site 0801), Montería
- Czechia (7):
  - FN Brno. ( Site 1501), Brno
  - Nemocnice Novy Jicin a.s. Clen skupiny AGEL ( Site 1506), Nový Jičín
  - Fakultni nemocnice Olomouc ( Site 1502), Olomouc
  - Fakultni nemocnice Ostrava ( Site 1507), Ostrava
  - Thomayerova nemocnice ( Site 1505), Prague
  - Fakultni nemocnice v Motole ( Site 1504), Prague
  - Nemocnice Na Bulovce ( Site 1503), Prague
- Finland (5):
  - HYKS ( Site 2300), Helsinki
  - Keski-Suomen keskussairaala ( Site 2303), Jyväskylä
  - Oulun yliopistollinen sairaala - OYS ( Site 2304), Oulu
  - TAYS ( Site 2301), Tampere
  - TYKS ( Site 2302), Turku
- France (11):
  - ICO Centre Paul Papin ( Site 2208), Angers
  - CHU Besancon - Hopital Jean Minjoz ( Site 2200), Besançon
  - Hopital Saint Andre ( Site 2202), Bordeaux
  - Hopital La Timone ( Site 2204), Marseille
  - CHU Saint-Eloi ( Site 2203), Montpellier
  - Centre Antoine Lacassagne ( Site 2211), Nice
  - Hopital Europeen Georges Pompidou ( Site 2206), Paris
  - Hospices Civils de Lyon Centre Hospitalier Lyon Sud ( Site 2212), Pierre-Bénite
  - Centre Eugene Marquis ( Site 2209), Rennes
  - Centre Rene Gauducheau ICO ( Site 2207), Saint-Herblain
  - Institut Claudius Regaud IUCT Oncopole ( Site 2201), Toulouse
- Germany (16):
  - Campus Charite Mitte ( Site 2120), Berlin
  - Helios Klinikum Berlin Buch ( Site 2125), Berlin
  - Universitaetsklinikum Bonn ( Site 2110), Bonn
  - Universitaetsklinikum der Technischen Universitaet Dresden ( Site 2113), Dresden
  - Universitatsklinikum Dusseldorf ( Site 2108), Düsseldorf
  - Universitaetsklinikum Erlangen. Waldkrankenhaus ( Site 2102), Erlangen
  - Universitaetsklinikum Essen ( Site 2116), Essen
  - Universitaetsklinikum Frankfurt ( Site 2121), Frankfurt
  - Universitaetsklinikum Freiburg ( Site 2119), Freiburg im Breisgau
  - Universitaetsklinikum Hamburg-Eppendorf ( Site 2118), Hamburg
  - Universitaetsklinikum Jena. ( Site 2104), Jena
  - Universitaetsklinikum Schleswig Holstein ( Site 2109), Lübeck
  - Universitaetsmedizin der Johannes Gutenberg-Universitaet Mainz ( Site 2111), Mainz
  - Studienpraxis Urologie ( Site 2115), Nürtingen
  - Krankenhaus der Barmherzigen Brueder Trier ( Site 2117), Trier
  - Universitaetsklinikum Tuebingen ( Site 2100), Tübingen
- Ireland (3):
  - Beaumont Hospital ( Site 1611), Dublin
  - St Vincents University Hospital ( Site 1610), Dublin
  - University Hospital Waterford ( Site 1614), Waterford
- Italy (8):
  - Ospedale San Luigi Gonzaga ( Site 2010), Orbassano, Torino
  - Medical Oncology Ospedale San Donato ( Site 2004), Arezzo
  - Istituto Scientifico Romagnolo per Studio e Cura Tumori IRST ( Site 2012), Meldola
  - Fondazione IRCCS Istituto Nazionale dei Tumori di Milano ( Site 2005), Milan
  - Istituto Europeo di Oncologia ( Site 2000), Milan
  - Azienda Ospedaliero Universitaria di Modena Policlinico ( Site 2006), Modena
  - Istituto Nazionale Tumori IRCCS Fondazione Pascale ( Site 2003), Napoli
  - Istituto Nazionale Tumori Regina Elena ( Site 2009), Roma
- Japan (21):
  - Nagoya University Hospital ( Site 0431), Nagoya, Aichi-ken
  - Sapporo Medical University Hospital ( Site 0424), Sapporo, Hokkaido
  - Kagawa University Hospital ( Site 0419), Kita-gun, Kagawa-ken
  - Japan Community Health care Organization Sendai Hospital ( Site 0430), Sendai, Miyagi
  - Nara Medical University Hospital ( Site 0416), Kashihara, Nara
  - Osaka Rosai Hospital ( Site 0418), Sakai, Osaka
  - Kindai University Hospital ( Site 0411), Sayama, Osaka
  - Saitama Medical University International Medical Center ( Site 0404), Hidaka, Saitama
  - Yamaguchi University Hospital ( Site 0406), Ube, Yamaguchi
  - Akita University Hospital ( Site 0433), Akita
  - Harasanshin Hospital ( Site 0402), Fukuoka
  - Kyushu University Hospital ( Site 0413), Fukuoka
  - Kumamoto University Hospital ( Site 0434), Kumamoto
  - Nagano Municipal Hospital ( Site 0429), Nagano
  - Niigata University Medical & Dental Hospital ( Site 0421), Niigata
  - Osaka International Cancer Institute ( Site 0401), Osaka
  - Osaka City University Hospital ( Site 0428), Osaka
  - Toranomon Hospital ( Site 0426), Tokyo
  - Nippon Medical School Hospital ( Site 0400), Tokyo
  - Keio University Hospital ( Site 0407), Tokyo
  - Toyama University Hospital ( Site 0432), Toyama
- Netherlands (3):
  - Amphia Ziekenhuis Breda ( Site 1901), Breda
  - Maastricht Universitair Medisch Centrum - MUMC ( Site 1902), Maastricht
  - Franciscus Gasthuis ( Site 1903), Rotterdam
- Poland (15):
  - Mazowiecki Szpital Onkologiczny ( Site 1316), Wieliszew, Masovian Voivodeship
  - Szpital Specjalistyczny w Koscierzynie Sp. z o.o. ( Site 1322), Kościerzyna, Pomeranian Voivodeship
  - Szpital Specjalistyczny w Brzozowie Podkarpacki Osrodek Onkologiczny ( Site 1309), Brzozów
  - Wojewodzki Szpital Specjalistyczny nr 4 w Bytomiu ( Site 1307), Bytom
  - Wojewodzkie Centrum Onkologii Copernicus ( Site 1304), Gdansk
  - Szpital Morski im. PCK Szpitale Wojewodzkie w Gdyni Sp. z o.o. ( Site 1302), Gdynia
  - Centrum Onkologii Instytut im. Marii Skłodowskiej Curie ( Site 1323), Gliwice
  - Przychodnia Lekarska Komed ( Site 1306), Konin
  - Centrum Onkologii Instytut im. Marii Sklodowskiej Curie ( Site 1310), Krakow
  - Centrum Onkologii Ziemi Lubelskiej im. sw. Jana z Dukli ( Site 1315), Lublin
  - Europejskie Centrum Zdrowia Otwock Szpital im. Fryderyka Chopina ( Site 1324), Otwock
  - Szpital Kliniczny Przemienienia Panskiego UM im. K. Marcinkowskiego ( Site 1311), Poznan
  - Wojewodzki Szpital Zespolony im. L. Rydygiera w Toruniu ( Site 1305), Torun
  - Centrum Medyczne Onkologii I Hipertermii ( Site 1321), Warsaw
  - Wojskowy Instytut Medyczny Centralny Szpital Medyczny MON ( Site 1300), Warsaw
- Russia (11):
  - Ivanovo Regional Oncology Dispensary ( Site 1204), Ivanovo
  - Krasnoyarsk Regional Clinical Oncological Dispensary ( Site 1210), Krasnoyarsk
  - N.N. Blokhin NMRCO ( Site 1206), Moscow
  - Russian Scientific Center of Roentgenoradiology ( Site 1201), Moscow
  - National Medical Research Radiology Centre ( Site 1200), Moscow
  - Bayandin Murmansk Regional Clinical Hospital ( Site 1214), Murmansk
  - Omsk Clinical Oncology Dispensary ( Site 1209), Omsk
  - Russian Scientific Center of Radiology and Surgical Technologies ( Site 1205), Saint Petersburg
  - Tomsk Scientific Research Institute of Oncology ( Site 1208), Tomsk
  - Republican Clinical Oncology Dispensary of Republic of Bashkortostan ( Site 1217), Ufa
  - Clinical Hospital Bashkirsky Medical State University ( Site 1202), Ufa
- South Korea (5):
  - National Cancer Center ( Site 0304), Goyang-si, Gyeonggi-do
  - Seoul National University Hospital ( Site 0302), Seoul
  - Severance Hospital Yonsei University Health System ( Site 0303), Seoul
  - Asan Medical Center ( Site 0300), Seoul
  - Samsung Medical Center ( Site 0301), Seoul
- Spain (9):
  - Hospital Universitario Infanta Cristina ( Site 1805), Badajoz
  - Hospital de la Santa Creu i Sant Pau ( Site 1807), Barcelona
  - Hospital de Girona Dr. Josep Trueta ( Site 1806), Girona
  - Hospital Universitario Gregorio Maranon ( Site 1801), Madrid
  - Hospital Universitario Ramon y Cajal ( Site 1800), Madrid
  - Hospital Universitario Virgen de la Victoria ( Site 1808), Málaga
  - Clinica Universitaria de Navarra ( Site 1803), Pamplona
  - Instituto Valenciano de Oncologia ( Site 1804), Valencia
  - Hospital Universitario y Politecnico La Fe de Valencia ( Site 1809), Valencia
- Taiwan (5):
  - China Medical University Hospital ( Site 0200), Taichung
  - Taichung Veterans General Hospital ( Site 0204), Taichung
  - National Taiwan University Hospital ( Site 0202), Taipei
  - Taipei Veterans General Hospital ( Site 0201), Taipei
  - Chang Gung Medical Foundation. Linkou ( Site 0203), Taoyuan District
- United Kingdom (8):
  - North Staffordshire Hospital in Stoke-on-Trent ( Site 1601), Stoke-on-Trent, Staffordshire
  - Western General Hospital ( Site 1600), Edinburgh
  - The Beatson West of Scotland Cancer Centre ( Site 1605), Glasgow
  - Royal Free Hospital ( Site 1609), London
  - St George s Healthcare Trust ( Site 1608), London
  - Charing Cross Hospital ( Site 1607), London
  - The Christie NHS Foundation Trust ( Site 1602), Manchester
  - The James Cook University Hospital ( Site 1606), Middlesbrough

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Choueiri TK, Tomczak P, Park SH, Venugopal B, Ferguson T, Symeonides SN, Hajek J, Chang YH, Lee JL, Sarwar N, Haas NB, Gurney H, Sawrycki P, Mahave M, Gross-Goupil M, Zhang T, Burke JM, Doshi G, Melichar B, Kopyltsov E, Alva A, Oudard S, Topart D, Hammers H, Kitamura H, McDermott DF, Silva A, Winquist E, Cornell J, Elfiky A, Burgents JE, Perini RF, Powles T; KEYNOTE-564 Investigators. Overall Survival with Adjuvant Pembrolizumab in Renal-Cell Carcinoma. N Engl J Med. 2024 Apr 18;390(15):1359-1371. doi: 10.1056/NEJMoa2312695. PMID 38631003
- [Derived] Choueiri TK, Tomczak P, Park SH, Venugopal B, Symeonides S, Hajek J, Ferguson T, Chang YH, Lee JL, Haas N, Sawrycki P, Sarwar N, Gross-Goupil M, Thiery-Vuillemin A, Mahave M, Kimura G, Perini RF, Saretsky TL, Bhattacharya R, Xu L, Powles T. Patient-Reported Outcomes in KEYNOTE-564: Adjuvant Pembrolizumab Versus Placebo for Renal Cell Carcinoma. Oncologist. 2024 Feb 2;29(2):142-150. doi: 10.1093/oncolo/oyad231. PMID 37589219
- [Derived] Powles T, Tomczak P, Park SH, Venugopal B, Ferguson T, Symeonides SN, Hajek J, Gurney H, Chang YH, Lee JL, Sarwar N, Thiery-Vuillemin A, Gross-Goupil M, Mahave M, Haas NB, Sawrycki P, Burgents JE, Xu L, Imai K, Quinn DI, Choueiri TK; KEYNOTE-564 Investigators. Pembrolizumab versus placebo as post-nephrectomy adjuvant therapy for clear cell renal cell carcinoma (KEYNOTE-564): 30-month follow-up analysis of a multicentre, randomised, double-blind, placebo-controlled, phase 3 trial. Lancet Oncol. 2022 Sep;23(9):1133-1144. doi: 10.1016/S1470-2045(22)00487-9. PMID 36055304
- [Derived] Choueiri TK, Tomczak P, Park SH, Venugopal B, Ferguson T, Chang YH, Hajek J, Symeonides SN, Lee JL, Sarwar N, Thiery-Vuillemin A, Gross-Goupil M, Mahave M, Haas NB, Sawrycki P, Gurney H, Chevreau C, Melichar B, Kopyltsov E, Alva A, Burke JM, Doshi G, Topart D, Oudard S, Hammers H, Kitamura H, Bedke J, Perini RF, Zhang P, Imai K, Willemann-Rogerio J, Quinn DI, Powles T; KEYNOTE-564 Investigators. Adjuvant Pembrolizumab after Nephrectomy in Renal-Cell Carcinoma. N Engl J Med. 2021 Aug 19;385(8):683-694. doi: 10.1056/NEJMoa2106391. PMID 34407342
- [Derived] Marconi L, Sun M, Beisland C, Klatte T, Ljungberg B, Stewart GD, Dabestani S, Choueiri TK, Bex A. Prevalence, Disease-free, and Overall Survival of Contemporary Patients With Renal Cell Carcinoma Eligible for Adjuvant Checkpoint Inhibitor Trials. Clin Genitourin Cancer. 2021 Apr;19(2):e92-e99. doi: 10.1016/j.clgc.2020.12.005. Epub 2021 Jan 7. PMID 33526329
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com/
- See also: Plain Language Summary — https://msd.trialsummaries.com/Study/StudyDetails?id=26135&tenant=MT_MSD_9011

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of the 994 participants randomized in the study, 984 participants received study medication and were evaluable for safety analyses (Database cutoff date 14 Dec 2020)
Groups:
- Pembrolizumab: Participants received pembrolizumab 200 mg via intravenous (IV) infusion on Day 1 of each 3-week cycle for up to 17 cycles (up to approximately 1 year).
- Placebo: Participants received placebo (saline solution) via IV infusion on Day 1 of each 3-week cycle for up to 17 cycles (up to approximately 1 year).
Period: Overall Study
Arm/Group | Pembrolizumab | Placebo
Started | 496 | 498
Treated | 488 | 496
Continuing Study Treatment | 0 | 1
Completed Study Treatment | 298 | 365
Discontinued Study Treatment | 190 | 130
Completed (Completed Trial) | 0 | 0
Not Completed | 496 | 498
Not completed — Death | 18 | 33
Not completed — Withdrawal by Subject | 15 | 11
Not completed — Ongoing on trial follow up | 463 | 454

BASELINE CHARACTERISTICS:
Population: All randomized participants
Groups:
- Total: Total of all reporting groups
Arm/Group | Pembrolizumab | Placebo | Total
Number analyzed (Participants) | 496 | 498 | 994
Age, Continuous [Mean (Standard Deviation); unit: Years] | 58.3 (10.6) | 58.6 (11.0) | 58.4 (10.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 149 | 139 | 288
  Male | 347 | 359 | 706
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 72 | 62 | 134
  Not Hispanic or Latino | 381 | 394 | 775
  Unknown or Not Reported | 43 | 42 | 85
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 10 | 2 | 12
  Asian | 63 | 75 | 138
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 7 | 5 | 12
  White | 372 | 377 | 749
  More than one race | 8 | 5 | 13
  Unknown or Not Reported | 36 | 34 | 70

OUTCOME MEASURES:

1. Primary Outcome: Disease-free Survival (DFS) as Assessed by the Investigator
Description: DFS, as assessed by the investigator, is defined as the time from randomization to the first documented local recurrence, distant kidney cancer metastasis(es), or death due to any cause, whichever occurs first. Cox regression model with Efron's method of tie handling with treatment as a covariate stratified by metastasis status (M0 versus M1 no evidence of disease (NED) by investigator) and Eastern Cooperative Oncology Group Performance Status (ECOG PS) (0 versus 1), United States (US) participant (Yes versus No) within M0 group by investigator was used to report hazard ratio (HR) and 95% confidence intervals (CIs).
Time Frame: Up to approximately 42 months (database cutoff date 14 Dec 2020)
Population: All randomized participants
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab | Placebo
Number analyzed (Participants) | 496 | 498
Months | NA [NA to NA] — NA = Median, lower and upper limit of 95% CIs for DFS was not reportable at the time of last disease assessment due to insufficient number of participants with events by the time of the data cutoff (14-Dec-2020). | NA [NA to NA] — NA = Median, lower and upper limit of 95% CIs for DFS was not reportable at the time of last disease assessment due to insufficient number of participants with events by the time of the data cutoff (14-Dec-2020).
Statistical Analysis 1: Comparison: Pembrolizumab vs Placebo; Test type: Other — HR and the associated 95% CIs were calculated based on Cox Regression model and p-value was calculated based on log-rank test, in accordance with the statistical analysis plan; p = 0.0010, Log Rank; One-sided p-value was based on log-rank test stratified by metastasis status, ECOG PS, US participant within M0 group by investigator; Hazard Ratio (HR) = 0.68, 95% CI 2-sided [0.53 to 0.87] — Cox regression model with Efron's method of tie handling with treatment as a covariate stratified by metastasis status, ECOG PS, and US participant within M0 group by investigator was used to calculate HR and 95% CIs

2. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the time from randomization to death due to any cause.
Time Frame: Up to approximately 72 months
Reporting Status: Not Posted, anticipated posting 2026-12

3. Secondary Outcome: Number of Participants Who Experienced an Adverse Event (AE)
Description: An AE is defined as any unfavorable and unintended change in the structure, function, or chemistry of the body temporally associated with the use of the study treatment, whether or not considered related to the use of study treatment. Participants are monitored for the occurrence of nonserious AEs for up to 30 days after last dose of study treatment and of serious AEs for up to 90 days after last dose of study treatment. The number of participants who experience an AE will be assessed.
Time Frame: Nonserious AEs: Up to 30 days after last dose of study treatment (Up to approximately 13 months); Serious AEs: Up to 90 days after last dose of study treatment (Up to approximately 15 months)
Reporting Status: Not Posted, anticipated posting 2026-12

4. Secondary Outcome: Number of Participants Who Discontinued Study Drug Due to an AE
Description: An AE is defined as any unfavorable and unintended change in the structure, function, or chemistry of the body temporally associated with the use of the study treatment, whether or not considered related to the use of study treatment. The number of participants who discontinue study treatment due to an AE will be assessed.
Time Frame: Up to approximately 12 months
Reporting Status: Not Posted, anticipated posting 2026-12

5. Secondary Outcome: First Local Disease Recurrence-specific Survival (DRSS1) as Assessed by the Investigator
Description: DRSS1 is defined as the time from randomization to the first documented local recurrence of RCC as assessed by the investigator. For DRSS1, only local recurrence is counted as an event.
Time Frame: Up to approximately 72 months
Reporting Status: Not Posted, anticipated posting 2026-12

6. Secondary Outcome: Second Disease Recurrence-Specific Survival (DRSS2) as Assessed by the Investigator
Description: DRSS2 is defined as the time from randomization to the first documented local recurrence with visceral lesion or occurrence of distant kidney cancer metastasis(es) with visceral lesion, whichever occurs first, as assessed by the investigator.
Time Frame: Up to approximately 72 months
Reporting Status: Not Posted, anticipated posting 2026-12

7. Secondary Outcome: Event-Free Survival (EFS) as Assessed by the Blinded Independent Central Review (BICR)
Description: EFS is defined as time from randomization to the first documented local recurrence or occurrence of distant kidney cancer metastasis(es) among participants which by BICR were considered disease-free at baseline (M0/M1 NED); or disease progression among participants which by BICR were considered to have baseline disease (M1), or death due to any cause, whichever occurs first.
Time Frame: Up to approximately 72 months
Reporting Status: Not Posted, anticipated posting 2026-12

8. Secondary Outcome: DFS According to Participant Programmed Cell Death-Ligand 1 (PD-L1) Expression Status (Positive, Negative) as Assessed by the Investigator
Description: DFS, as assessed by the investigator, is defined as the time from randomization to the first documented local recurrence, or occurrence of distant kidney cancer metastasis(es), or death due to any cause, whichever occurs first. The PD-L1 expression status is based on combined positive score (CPS). If CPS is ≥ 1, PD-L1 expression status is positive and if the CPS is <1, PD-L1 expression status is negative.
Time Frame: Up to approximately 72 months
Reporting Status: Not Posted, anticipated posting 2026-12

9. Secondary Outcome: OS According to Participant PD-L1 Expression Status (Positive, Negative)
Description: OS is defined as the time from randomization to death due to any cause. The PD-L1 expression status is based on combined positive score (CPS). If CPS is ≥ 1, PD-L1 expression status is positive and if the CPS is <1, PD-L1 expression status is negative.
Time Frame: Up to approximately 72 months
Reporting Status: Not Posted, anticipated posting 2026-12

10. Secondary Outcome: Change From Baseline in the European Organization for the Research and Treatment of Cancer Quality of Life Questionnaire C30 (EORTC QLQ-C30) Total Score
Description: The QLQ-C30 quality of life (QOL) questionnaire contains 5 functioning scales (physical, role, cognitive, emotional, and social), 3 symptom scales (fatigue, nausea and vomiting, and pain) and single symptom items (dyspnoea, loss of appetite, insomnia, constipation and diarrhoea) and perceived financial impact of the disease. Items are scored on a 4-point scale (1=not at all, 2=a little, 3= quite a bit, 4=very much). The QLQC30 also contains 2 global health status scales that use 7-point scale scoring (1=very poor and 7=excellent). The change from baseline in the 2-item global health status/QOL life scale (range: 2-14) will be presented, with a higher score representing a higher QOL.
Time Frame: Baseline and Week 52
Reporting Status: Not Posted, anticipated posting 2026-12

11. Secondary Outcome: Change From Baseline in the Functional Assessment of Cancer Therapy Kidney Symptom Index-Disease Related Symptoms (FKSI-DRS) Index Score
Description: The FKSI-DRS index consists of a 9-item questionnaire that assesses the extent of participant symptoms from kidney cancer over the previous 7 days. Responses are scored on a 5-point scale (0=Not at all to 4=Very much) and summed to generate an index symptom score. These scores can range from 0 to 36, with a higher score indicating more favorable kidney cancer symptom status. The change from baseline in the FKSI-DRS index score will be presented.
Time Frame: Baseline and Week 52
Reporting Status: Not Posted, anticipated posting 2026-12

ADVERSE EVENTS:
Time Frame: Up to approximately 43 months (Database cutoff date 14 Dec 2020).
Description: All-cause mortality was reported on all randomized participants. Serious and non-serious AEs were reported among participants who received at least one dose of study treatment.
Arm/Group | Pembrolizumab | Placebo
All-Cause Mortality (participants affected / at risk) | 18/496 | 33/498
Serious Adverse Events (participants affected / at risk) | 100/488 | 56/496
Other Adverse Events (participants affected / at risk) | 436/488 | 393/496
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pembrolizumab (N=488) | Placebo (N=496)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 2 (2) | 2 (2)
Bundle branch block left (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure (Cardiac disorders) | 2 (2) | 1 (1)
Coronary artery stenosis (Cardiac disorders) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 3 (3) | 0 (0)
Myocarditis (Cardiac disorders) | 1 (1) | 0 (0)
Pleuropericarditis (Cardiac disorders) | 1 (2) | 0 (0)
Sinus node dysfunction (Cardiac disorders) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Adrenal insufficiency (Endocrine disorders) | 6 (6) | 0 (0)
Autoimmune thyroiditis (Endocrine disorders) | 1 (1) | 0 (0)
Glucocorticoid deficiency (Endocrine disorders) | 1 (1) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 2 (2) | 0 (0)
Hypophysitis (Endocrine disorders) | 1 (1) | 0 (0)
Thyroiditis (Endocrine disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 1 (1)
Abdominal wall haematoma (Gastrointestinal disorders) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 5 (5) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diverticulum (Gastrointestinal disorders) | 1 (1) | 0 (0)
Enterocolitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
Large intestine polyp (Gastrointestinal disorders) | 0 (0) | 1 (1)
Mallory-Weiss syndrome (Gastrointestinal disorders) | 0 (0) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (2) | 0 (0)
Influenza like illness (General disorders) | 1 (1) | 0 (0)
Multiple organ dysfunction syndrome (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cholestasis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatitis (Hepatobiliary disorders) | 2 (2) | 0 (0)
Hepatitis alcoholic (Hepatobiliary disorders) | 0 (0) | 1 (1)
Immune-mediated hepatitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Anorectal infection (Infections and infestations) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0)
Campylobacter infection (Infections and infestations) | 0 (0) | 1 (1)
Device related infection (Infections and infestations) | 0 (0) | 1 (2)
Encephalitis (Infections and infestations) | 1 (1) | 0 (0)
Helicobacter infection (Infections and infestations) | 0 (0) | 1 (1)
Infected lymphocele (Infections and infestations) | 0 (0) | 1 (1)
Infection (Infections and infestations) | 1 (2) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 0 (0)
Intervertebral discitis (Infections and infestations) | 0 (0) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 2 (2) | 0 (0)
Meningitis aseptic (Infections and infestations) | 2 (2) | 0 (0)
Pneumonia (Infections and infestations) | 6 (6) | 1 (1)
Pneumonia influenzal (Infections and infestations) | 0 (0) | 1 (1)
Pyelonephritis (Infections and infestations) | 1 (1) | 0 (0)
Rectal abscess (Infections and infestations) | 0 (0) | 1 (1)
Respiratory tract infection (Infections and infestations) | 2 (2) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 1 (1)
Septic shock (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 2 (2)
Vascular device infection (Infections and infestations) | 0 (0) | 1 (1)
Viral infection (Infections and infestations) | 1 (1) | 1 (1)
Wound infection (Infections and infestations) | 1 (1) | 1 (1)
Accidental overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Craniocerebral injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Incisional hernia (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Infusion related reaction (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Joint dislocation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Multiple injuries (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Nail injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post procedural haematuria (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Tendon rupture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 5 (6) | 0 (0)
Glucose tolerance impaired (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperamylasaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 4 (4) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Chondrocalcinosis pyrophosphate (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Sjogren's syndrome (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Trigger finger (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 3 (3)
Basal cell carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Benign lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Choroid melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Colon neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Neuroendocrine tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Primary myelofibrosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Ataxia (Nervous system disorders) | 0 (0) | 1 (1)
Cerebellar ischaemia (Nervous system disorders) | 1 (1) | 0 (0)
Cerebellar syndrome (Nervous system disorders) | 1 (1) | 0 (0)
Cerebral infarction (Nervous system disorders) | 1 (1) | 0 (0)
Cerebral ischaemia (Nervous system disorders) | 1 (2) | 0 (0)
Cognitive disorder (Nervous system disorders) | 1 (1) | 0 (0)
Facial paralysis (Nervous system disorders) | 1 (1) | 0 (0)
Haemorrhage intracranial (Nervous system disorders) | 0 (0) | 1 (1)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 2 (2)
Loss of consciousness (Nervous system disorders) | 1 (1) | 0 (0)
Myasthenic syndrome (Nervous system disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 2 (2)
Tension headache (Nervous system disorders) | 1 (1) | 0 (0)
Transient global amnesia (Nervous system disorders) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 1 (1)
Suicide attempt (Psychiatric disorders) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 6 (6) | 0 (0)
Bladder mass (Renal and urinary disorders) | 1 (1) | 0 (0)
Calculus urinary (Renal and urinary disorders) | 0 (0) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 2 (3)
Renal colic (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal pain (Renal and urinary disorders) | 0 (0) | 1 (1)
Tubulointerstitial nephritis (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 1 (1) | 2 (2)
Testicular torsion (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Uterine polyp (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Immune-mediated pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3)
Lichenification (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Stevens-Johnson syndrome (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Essential hypertension (Vascular disorders) | 1 (1) | 0 (0)
Giant cell arteritis (Vascular disorders) | 1 (1) | 0 (0)
Haematoma (Vascular disorders) | 0 (0) | 1 (1)
Orthostatic hypotension (Vascular disorders) | 1 (1) | 0 (0)
Vasculitis (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pembrolizumab (N=488) | Placebo (N=496)
Hyperthyroidism (Endocrine disorders) | 56 (58) | 1 (1)
Hypothyroidism (Endocrine disorders) | 103 (111) | 18 (20)
Abdominal pain (Gastrointestinal disorders) | 36 (54) | 39 (50)
Constipation (Gastrointestinal disorders) | 35 (39) | 40 (42)
Diarrhoea (Gastrointestinal disorders) | 123 (195) | 111 (171)
Dry mouth (Gastrointestinal disorders) | 33 (37) | 5 (5)
Nausea (Gastrointestinal disorders) | 80 (105) | 48 (61)
Vomiting (Gastrointestinal disorders) | 39 (44) | 28 (31)
Asthenia (General disorders) | 50 (85) | 36 (50)
Fatigue (General disorders) | 145 (180) | 120 (156)
Influenza like illness (General disorders) | 25 (26) | 21 (24)
Oedema peripheral (General disorders) | 21 (26) | 27 (30)
Pyrexia (General disorders) | 31 (31) | 22 (24)
Nasopharyngitis (Infections and infestations) | 28 (33) | 42 (47)
Upper respiratory tract infection (Infections and infestations) | 27 (32) | 24 (27)
Urinary tract infection (Infections and infestations) | 29 (36) | 20 (30)
Alanine aminotransferase increased (Investigations) | 35 (42) | 17 (23)
Aspartate aminotransferase increased (Investigations) | 36 (40) | 10 (14)
Blood creatinine increased (Investigations) | 50 (59) | 42 (52)
Decreased appetite (Metabolism and nutrition disorders) | 34 (34) | 10 (10)
Hyperglycaemia (Metabolism and nutrition disorders) | 28 (36) | 17 (20)
Arthralgia (Musculoskeletal and connective tissue disorders) | 108 (159) | 93 (123)
Back pain (Musculoskeletal and connective tissue disorders) | 49 (56) | 63 (70)
Myalgia (Musculoskeletal and connective tissue disorders) | 46 (60) | 32 (38)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 35 (41) | 25 (30)
Dizziness (Nervous system disorders) | 39 (47) | 27 (32)
Headache (Nervous system disorders) | 69 (92) | 62 (91)
Insomnia (Psychiatric disorders) | 26 (27) | 29 (32)
Cough (Respiratory, thoracic and mediastinal disorders) | 76 (90) | 50 (56)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 30 (32) | 27 (38)
Dry skin (Skin and subcutaneous tissue disorders) | 26 (30) | 22 (22)
Pruritus (Skin and subcutaneous tissue disorders) | 111 (148) | 65 (75)
Rash (Skin and subcutaneous tissue disorders) | 98 (151) | 53 (83)
Hypertension (Vascular disorders) | 38 (46) | 39 (43)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator agrees to submit all manuscripts or abstracts to the sponsor before submission. This allows the sponsor to protect proprietary information and to provide comments.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-10-13): https://cdn.clinicaltrials.gov/large-docs/34/NCT03142334/Prot_SAP_000.pdf